CLINICAL TRIAL: NCT04182204
Title: A Phase III, Open-Label, Multicenter, Randomized, Study Evaluating the Safety and Efficacy of Polatuzumab Vedotin in Combination With Rituximab Plus Gemcitabine Plus Oxaliplatin (R-GEMOX) Versus R-GEMOX Alone in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study to Evaluate the Safety and Efficacy of Polatuzumab Vedotin in Combination With Rituximab, Gemcitabine and Oxaliplatin Compared to Rituximab, Gemcitabine and Oxaliplatin Alone in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: POLARGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO40598; 2018-003727-10 (EudraCT Number)
Record Dates: First submitted 2019-11-18; First posted 2019-12-02 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma; Large B-Cell; Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — polatuzumab vedotin; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: In stage 1 participants are all assigned to one group. In stage 2 participants are assigned to two groups in parallel for the duration of the study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pola-R-GemOx (Stage 1) (Experimental): Participants will receive polatuzumab vedotin 1.8 milligrams per kilogram (mg/kg) for a maximum dose of 240 mg per cycle (mg/cycle) administered intravenously (IV) and rituximab 375 milligrams per square meter (mg/m^2) administered IV on Day 1. Participants will receive gemcitabine 1000 mg/m^2 administered IV and oxaliplatin 100 mg/m^2 administered IV on Day 2. Each cycle will consist of 21 days with up to 8 cycles of treatment administration.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin
- Pola-R-GemOx (Stage 2) (Experimental): Participants will receive polatuzumab vedotin 1.8 mg/kg for a maximum dose of 240 mg/cycle administered IV and rituximab 375 mg/m^2 administered IV on Day 1. Participants will receive gemcitabine 1000 mg/m^2 administered IV and oxaliplatin 100 mg/m^2 administered IV on Day 2. Each cycle will consist of 21 days with up to 8 cycles of treatment administration.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin
- R-GemOx (Stage 2) (Active Comparator): Participants will receive rituximab 375 mg/m^2 administered IV on Day 1. Participants will receive gemcitabine 1000 mg/m^2 administered IV and oxaliplatin 100 mg/m^2 administered IV on Day 2. Each cycle will consist of 21 days with up to 8 cycles of treatment administration.
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin 1.8 mg/kg for a maximum dose of 240 mg/cycle IV on Day 1 of each 21-day cycle for up to 8 cycles.
  Arms: Pola-R-GemOx (Stage 1); Pola-R-GemOx (Stage 2)
Drug: Rituximab — Rituximab 375 mg/m2 IV on Day 1 of each 21-day cycle for up to 8 cycles.
  Other Names: Mabthera; Rituxan
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV on Day 2 of each 21-day cycle for up to 8 cycles.
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 IV on Day 2 of each 21-day cycle for up to 8 cycle.

SUMMARY:
This study is a multicenter, open-label study of polatuzumab vedotin administered by intravenous (IV) infusion in combination with rituximab, gemcitabine and oxaliplatin (R-GemOx) in participants with relapsed or refractory diffuse large B-cell lymphoma (DLBCL). The study comprises of two stages: a safety run-in stage and a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The safety run-in stage (Stage 1) will assess the safety of polatuzumab vedotin plus rituximab, gemcitabine and oxaliplatin (Pola-R-GemOx) in 10 participants. The randomized controlled trial (RCT) (Stage 2) will compare Pola-R-GemOx versus R-GemOx alone using overall survival (OS). This is an event-driven trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diffuse large B-cell lymphoma, not otherwise specified (NOS) or history of transformation of indolent disease to DLBCL
* Relapsed disease (disease that has recurred following a response that lasted ≥ 6 months from completion of the last line of therapy) or refractory disease (disease that did not respond to or that progressed during therapy or progressed within 6 months (< 6 months) of prior therapy)
* At least one (≥ 1) line of prior systemic therapy:
* Patients may have undergone autologous hematopoietic stem cell transplantation (HSCT) prior to recruitment; In such cases, salvage chemotherapy (e.g., rituximab, dexamethasone, cytarabine, and cisplatin [R-DHAP] and rituximab, ifosfamide, carboplatin, and etoposide phosphate [R-ICE]) will be counted as one line of therapy and conditioning chemotherapy (e.g., BEAM) followed by consolidative autologous HSCT will be counted as one line of therapy
* Patients may have undergone allogeneic HSCT prior to recruitment, so long as they are off all immunosuppressive therapy and have no active GVHD; In such cases, salvage chemotherapy (e.g., R-DHAP and R-ICE) will be counted as one line of therapy and conditioning chemotherapy (e.g., carmustine, etoposide, cytarabine, and melphalan [BEAM]) followed by allogeneic HSCT will be counted as a separate line of therapy
* Participants may have undergone CAR T-cell therapy prior to recruitment. In such cases, cell collection, conditioning chemotherapy, and infusion will be counted as one line of therapy.
* Local therapies (e.g., radiotherapy) will not be considered as lines of treatment
* For participants with a history of the transformation of indolent disease to DLBCL, it is preferred that participants have received at least one treatment for the transformed lymphoma. However, if there are cases where the participants have received an anthracycline-containing chemotherapy regimen (such as R-CHOP) for the indolent lymphoma only, then these participants can be considered as eligible.
* At least one bi-dimensionally measurable lesion, defined as > 1.5 cm in its longest dimension as measured by CT or MRI
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
* Adequate hematological function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm,

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to rituximab, gemcitabine or oxaliplatin
* Peripheral neuropathy assessed to be > Grade 1 according to NCI CTCAE v5.0
* Prior use of polatuzumab vedotin or a gemcitabine plus platinum-based agent combination, recent participation in a clinical trial, and/or treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy within 2 weeks
* Planned autologous or allogenic stem cell transplantation or CAR T-cell therapy at time of recruitment
* Primary or secondary central nervous system (CNS) lymphoma
* Richter's transformation or prior CLL
* Abnormal laboratory values or health conditions, as assessed by the investigator, any known conditions preventing adherence to protocol or active bacterial, viral, fungal, mycobacterial, parasitic, or other infection
* Vaccination with a live vaccine within 4 weeks prior to treatment
* Recent major surgery (within 6 weeks before the start of Cycle 1 Day 1) other than for diagnosis
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 12 months after the last dose of study drug
* Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (7):
  - Cancer Specialists, Jacksonville, Florida
  - Memorial Cancer Institute at Memorial West, Pembroke Pines, Florida
  - IHA Hematology Oncology Consultants - Ann Arbor, Ann Arbor, Michigan
  - MSKCC at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Bergen, Montvale, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
- Brazil (4):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - Niagara Health Systems - St. Catherines General Site, St. Catharines, Ontario
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
- China (8):
  - Hu Nan Provincial Cancer Hospital, Changsha
  - West China Hospital - Sichuan University, Chengdu
  - Cancer Center, Sun Yat-sen University of Medical Sciences, Guangzhou
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Institute of Hematology and Hospital of Blood Disease, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- Finland (2):
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- France (5):
  - Hopital Henri Mondor, Créteil
  - Hopital De Haut Leveque, Pessac
  - Centre Henri Becquerel, Rouen
  - ICANS, Strasbourg
  - Hopital Bretonneau, Tours
- Universitätsklinikum Ulm, Ulm, Germany
- Greece (2):
  - Laiko General Hospital, Athens
  - Attiko Hospital, Athens
- India (3):
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - All India Institute of Medical Sciences ,Institute Rotary Cancer Hospital, New Delhi, National Capital Territory of Delhi
  - Tata Medical Center, Kolkata, West Bengal
- St James' Hospital, Dublin, Ireland
- Italy (4):
  - Uni Degli Studi Di Bari, Policlinico, Bari, Apulia
  - Azienda Ospedaliero-Universitaria Policlinico di Modena Ematologia, Modena, Emilia-Romagna
  - Az. Osp. Uni Ria Policlinico Tor Vergata, Rome, Lazio
  - USL 4 di Prato - Nuovo Ospeale di Prato, Prato, Tuscany
- Mexico (3):
  - Hospital de Especialidades Centro Medico Nacional La Raza, Mexico City, Mexico CITY (federal District)
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Cancerologia, Distrito Federal
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Gyeongsang National University Hospital, Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Univ. 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Dr. Peset, Valencia
- Turkey (Türkiye) (7):
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi, Adapazari/Sakarya
  - Abdurrahman Yurtarslan Onkoloji Training and Research Hospital, Ankara
  - Akdeniz Uni School of Medicine, Antalya
  - Istanbul Uni Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Amerikan HAstanesi Onkoloji Birimi Te?vikiye, Ni?anta??
- United Kingdom (2):
  - Kings College Hospital, London
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing/).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 270 participants with relapsed/refractory (r/r) diffuse large b-cell lymphoma (DLBCL) took part in the study at 64 investigative sites in 16 countries from 07 February 2020 to 29 November 2024.
Pre-assignment Details: The study was divided into 2 stages: Stage 1, or safety run-in (SRI), and Stage 2, or randomized controlled trial (RCT). Participants received polatuzumab vedotin in combination with rituximab + gemcitabine + oxaliplatin (Pola-R-GemOx) during the SRI stage. Participants were randomized in a 1:1 ratio to receive either Pola-R-GemOx or rituximab + gemcitabine + oxaliplatin (R-GemOx) in the RCT stage.
Groups:
- Stage 1: Pola-R-GemOx: Participants received rituximab, 375 milligrams per square meter (mg/m^2), intravenously (IV), followed by polatuzumab vedotin, 1.8 milligrams per kilogram (mg/kg), IV on Day 1 of each 21-day cycle. Participants also received gemcitabine, 1000 mg/m^2, IV followed by oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
- Stage 2: R-GemOx: Participants received rituximab, 375 mg/m^2, IV on Day 1, followed by gemcitabine, 1000 mg/m^2, IV and oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
- Stage 2: Pola-R-GemOx: Participants received rituximab, 375 mg/m^2, IV, followed by polatuzumab vedotin, 1.8 mg/kg, IV on Day 1 of each 21-day cycle. Participants also received gemcitabine, 1000 mg/m^2, IV followed by oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
Period: Safety Run-in
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Started | 15 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 10 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Death | 7 | 0 | 0
Period: Randomized Controlled Trial
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Started | 0 | 126 | 129
Safety-evaluable Population (Safety-evaluable population included all participants who received any amount of any study drug (regardless of the stage). One participant in the Pola-R-GemOx (randomized) arm and one participant in the R-GemOx (randomized) arm did not receive any treatment and were excluded from the safety-evaluable population.) | 0 | 125 | 128
Completed | 0 | 32 | 55
Not Completed | 0 | 94 | 74
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 10 | 6
Not completed — Death | 0 | 83 | 66

BASELINE CHARACTERISTICS:
Population: Enrolled population included all enrolled participants (regardless of the stage).
Groups:
- Stage 1: Pola-R-GemOx; Stage 2: Pola-R-GemOx: Participants received rituximab, 375 mg/m^2, IV, followed by polatuzumab vedotin, 1.8 mg/kg, IV on Day 1 of each 21-day cycle. Participants also received gemcitabine, 1000 mg/m^2, IV followed by oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
- Total: Total of all reporting groups
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx | Total
Number analyzed (Participants) | 15 | 126 | 129 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (12.6) | 62.2 (13.9) | 63.0 (14.5) | 63.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 65 | 56 | 128
  Male | 8 | 61 | 73 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 26 | 27 | 54
  Not Hispanic or Latino | 13 | 90 | 97 | 200
  Unknown or Not Reported | 1 | 10 | 5 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 9 | 7 | 16
  Asian | 1 | 41 | 49 | 91
  Black or African American | 0 | 6 | 3 | 9
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  White | 14 | 56 | 60 | 130
  Other | 0 | 6 | 8 | 14
  Multiple | 0 | 0 | 0 | 0
  Unknown | 0 | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From treatment initiation until 90 days after the last dose of study drug or initiation of non-protocol-specified anti-lymphoma treatment (NALT) (Up to approximately 8.3 months)
Population: Safety run-in population included all participants who received any amount of any study drug during safety run-in stage.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Pola-R-GemOx
Number analyzed (Participants) | 15
Participants | 14

2. Primary Outcome: Stage 1: Number of Participants With Peripheral Neuropathy (PN)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Participants receiving polatuzumab vedotin may develop PN, including peripheral sensory and/or motor neuropathy. Symptoms included hypoesthesia, hyperesthesia, paresthesia, dysesthesia, discomfort, a burning sensation, weakness, gait disturbance, loss of balance, orthostatic hypotension, syncope, or neuropathic pain.
Time Frame: From treatment initiation until 90 days after the last dose of study drug or initiation of NALT (Up to approximately 8.3 months)
Population: Safety run-in population included all participants who received any amount of any study drug during safety run-in stage.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Pola-R-GemOx
Number analyzed (Participants) | 15
Participants | 8

3. Primary Outcome: Stage 2: Overall Survival (OS)
Description: OS was defined as the time from randomization to the death from any cause during the study. Participants who were not reported as having died at the time of analysis were censored at the date when they were last known to be alive. Participants who did not have post-baseline information were censored at the date of randomization. Kaplan-Meier (KM) method was used to estimate median OS for each treatment arm.
Time Frame: From randomization to death (Up to approximately 34 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
months | 12.5 [8.9 to 15.8] | 19.5 [13.3 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; p = 0.0017, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.43 to 0.83]

4. Secondary Outcome: Stage 1 and Stage 2: Progression-free Survival (PFS)
Description: PFS=time from randomization to the first occurrence of disease progression (PD) (based on either: PET-CT data/not including any PET data), as determined by investigator, per Lugano response criteria or death due to any cause, whichever occurs first. PD based on PET-CT data=score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver &/or new lesions) on 5-point scale (5PS) with an increase in intensity of uptake from baseline at individual target nodes/nodal masses and/or new FDG-avid foci extranodal lesions consistent with lymphoma at interim or end-of-treatment assessment. New lesions: New FDG-avid foci consistent with lymphoma rather than another etiology, Bone marrow: New/recurrent FDG-avid foci. Participants who did not report PD nor died at time of analysis were censored on the date of last evaluable tumor assessment if post-baseline tumor assessment or on date of randomization if no post-baseline tumor assessment. KM methodology was used to estimate median PFS.
Time Frame: From randomization to first occurrence of PD or death (Up to approximately 34 months)
Population: Safety run-in population included all participants who received any amount of any study drug during stage 1. ITT population included all randomized participants in stage 2.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Stage 2: R-GemOx: R-GemOx: Participants received rituximab, 375 mg/m^2, IV on Day 1, followed by gemcitabine, 1000 mg/m^2, IV and oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
- Stage 2: Pola-R-GemOx: Participants received rituximab, 375 mg/m^2, IV, followed by polatuzumab vedotin,1.8 mg/kg, IV on Day 1 of each 21-day cycle. Participants also received gemcitabine, 1000 mg/m^2, IV followed by oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 126 | 129
months | 3.9 [3.0 to 6.3] | 2.7 [2.4 to 3.3] | 7.4 [6.2 to 11.7]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.27 to 0.51]

5. Secondary Outcome: Stage 2: Complete Response Rate (CRR), as Determined by an Independent Review Committee (IRC) at the End of Treatment
Description: CRR was defined as the percentage of participants who had a complete metabolic response (CMR) based on positron emission tomography-computed tomography (PET-CT) according to Lugano response criteria at the end of treatment as determined by IRC. CMR was defined as score 1, 2, or 3 (1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake >mediastinum but ≤ liver) with or without a residual mass on 5PS at lymph nodes and extra lymphatic sites. In Waldeyer's ring or extranodal sites with high physiologic uptake or with activation within spleen or marrow (e.g., with chemotherapy/myeloid colony-stimulating factors), uptake may be greater than normal mediastinum and/or liver. In this circumstance, CMR was inferred if uptake at sites of initial involvement was no greater than surrounding normal tissue even if the tissue had high physiologic uptake; no new lesions and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. Percentages are rounded off.
Time Frame: Up to approximately 8.5 months
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
percentage of participants | 19.0 [12.60 to 27.00] | 40.3 [31.77 to 49.30]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Response Rate = 21.26, 95% CI 2-sided [9.58 to 32.94]

6. Secondary Outcome: Stage 2: Objective Response Rate (ORR) as Determined by an IRC at End of Treatment
Description: ORR=percentage of participants with CMR/partial metabolic responses (PMR), based on PET-CT per Lugano response criteria as per an IRC. CMR=score 1, 2, or 3 with/ without a residual mass on 5PS at lymph nodes (LN) & extra lymphatic sites. In Waldeyer's ring or extra nodal sites with high physiologic uptake or with activation within spleen/marrow, uptake may be greater than normal mediastinum &/or liver. In this case, CMR was inferred if uptake at sites of initial involvement was no greater than surrounding normal tissue even if the tissue had high physiologic uptake; no new lesions & no evidence of FDG-avid disease in bone marrow. PMR=score 4 or 5 on 5PS (4=uptake moderately > liver; 5=uptake markedly higher than liver &/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size at LN & extra lymphatic sites; no new lesions & residual uptake higher than uptake in normal marrow but reduced compared with baseline. Percentages are rounded off.
Time Frame: Up to approximately 8.5 months
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
percentage of participants | 24.6 [17.37 to 33.07] | 52.7 [43.74 to 61.56]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Response Rate = 28.11, 95% CI 2-sided [15.89 to 40.33]

7. Secondary Outcome: Stage 1 and Stage 2: Percentage of Participants With Best Overall Response (BOR) as Determined by the Investigator
Description: BOR was defined as the best response while on study (based on PET-CT or CT data) according to Lugano response criteria, as determined by the investigator. CMR and PMR based on PET-CT data were defined as outlined in the ORR outcome measure (OM) number 8. CT-based complete radiologic response was defined as target lymphatic nodes/nodal masses regression to ≤ 1.5 centimeters (cm) in longest transverse diameter of a lesion (LDi); no extralymphatic sites of disease; absence of non-measured lesion; enlarged organs regress to normal; no new lesions and bone marrow normal by morphology, if indeterminate, immunohistochemistry (IHC) negative. CT-based partial response was defined as ≥50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of up to 6 target measurable nodes and extra nodal sites; absent/normal, regressed, but no increase in non-measured lesions; spleen regressed by >50% in length beyond normal and no new lesions. Percentages are rounded off.
Time Frame: Up to approximately 34 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 126 | 129
percentage of participants | 46.7 [21.27 to 73.41] | 34.9 [26.65 to 43.92] | 65.1 [56.23 to 73.29]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Difference in Response Rate = 30.20, 95% CI 2-sided [17.71 to 42.68]

8. Secondary Outcome: Stage 1 and Stage 2: CRR as Determined by the Investigator at End of Treatment
Description: CRR was defined as the percentage of participants who had CMR based positron emission tomography-computed tomography (PET-CT) according to Lugano response criteria at the end of treatment as determined by investigator. CMR was defined as score 1, 2, or 3 (1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake >mediastinum but ≤ liver) with or without a residual mass on 5PS at lymph nodes and extra lymphatic sites. In Waldeyer's ring or extranodal sites with high physiologic uptake or with activation within spleen or marrow (e.g., with chemotherapy/myeloid colony-stimulating factors), uptake may be greater than normal mediastinum and/or liver. In this circumstance, CMR was inferred if uptake at sites of initial involvement is no greater than surrounding normal tissue even if the tissue has high physiologic uptake; no new lesions and no evidence of FDG-avid disease in bone marrow. Percentages are rounded off.
Time Frame: Stage 1: Up to approximately 6.2 months and Stage 2: Up to approximately 8.5 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 126 | 129
percentage of participants | 20.0 [4.33 to 48.09] | 18.3 [11.94 to 26.12] | 35.7 [27.42 to 44.57]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Difference in Response Rate = 17.40, 95% CI 2-sided [5.95 to 28.86]

9. Secondary Outcome: Stage 1 and Stage 2: ORR as Determined by the Investigator at End of Treatment
Description: ORR=percentage of participants with CMR/PMR, based on PET-CT as determined by investigator per Lugano response criteria. CMR=score 1, 2, or 3 with/ without a residual mass on 5PS at LN & extra lymphatic sites. In Waldeyer's ring or extra nodal sites with high physiologic uptake or with activation within spleen/marrow, uptake may be greater than normal mediastinum &/or liver. In this case, CMR was inferred if uptake at sites of initial involvement was no greater than surrounding normal tissue even if the tissue had high physiologic uptake; no new lesions & no evidence of FDG-avid disease in bone marrow. PMR=score 4 or 5 on 5PS (4=uptake moderately > liver; 5=uptake markedly higher than liver &/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size at LN & extra lymphatic sites; no new lesions & residual uptake higher than uptake in normal marrow but reduced compared with baseline. Percentages are rounded off.
Time Frame: Stage 1: Up to approximately 6.2 months and Stage 2: Up to approximately 8.5 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 126 | 129
percentage of participants | 26.7 [7.79 to 55.10] | 24.6 [17.37 to 33.07] | 45.0 [36.20 to 53.96]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Difference in Response Rate = 20.36, 95% CI 2-sided [8.16 to 32.56]

10. Secondary Outcome: Stage 2: Duration of Response (DOR)
Description: DOR=time from the date of the first occurrence of a documented objective response (complete or partial response [CR/PR]) (based on PET-CT or CT data) as determined by the investigator, using Lugano response criteria, until PD (based on either response: including PET-CT data or not including any PET data) or death, whichever occurred first. CMR and PMR based on PET-CT data were defined as outlined in the ORR OM. CT-based complete and partial response were defined as outlined in the BOR OM. PD defined as outlined in the PFS OM.
Time Frame: Up to approximately 34 months
Population: DOR-evaluable population included all participants who had an objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 44 | 84
months | 8.5 [3.7 to 26.9] | 11.8 [8.6 to 15.5]

11. Secondary Outcome: Stage 1 and Stage 2: Event-free Survival (EFSeff)
Description: EFSeff was defined as the time from randomization to first to the earliest occurrence of the following: PD or relapse using Lugano response criteria (based on either response: including PET-CT data or not including any PET data); death due to any cause or initiation of any NALT. PD based on PET-CT data was defined as score 4 or 5 on 5PS with an increase in intensity of uptake from baseline at individual target nodes/nodal masses and/or new FDG-avid foci extranodal lesions consistent with lymphoma at interim or end-of-treatment assessment. New lesions: New FDG-avid foci consistent with lymphoma rather than another etiology, Bone marrow: New or recurrent FDG-avid foci. Participants with no EFSeff events were censored at the time of the last evaluable tumor assessment if post-baseline assessments were available and participants who did not undergo a post-baseline tumor assessment were censored at the time of randomization. KM method was used to estimate median EFS for each treatment arm.
Time Frame: Up to approximately 34 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 126 | 129
months | 3.9 [3.2 to 6.3] | 2.7 [2.5 to 3.3] | 6.8 [5.9 to 9.3]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.30 to 0.53]

12. Secondary Outcome: Stage 2: Time to Deterioration in Physical Functioning as Measured by the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire, Core 30 (EORTC QLQ-C30)
Description: Time to deterioration was defined as the time from randomization to the first documentation of a 10-point decrease in EORTC QLQ-C30 physical functioning scale. EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), global health status and quality of life (GHS/QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The functioning items were scored on a 4-point scale that ranged from "not at all" to "very much". Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher functioning). KM method was used to estimate median time to deterioration for each treatment arm.
Time Frame: Up to approximately 34 months
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
months | 2.8 [1.4 to 3.0] | 8.1 [4.2 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.40 to 0.83]

13. Secondary Outcome: Stage 2: Time to Deterioration in Fatigue Scale as Measured by the EORTC QLQ-C30
Description: Time to deterioration was defined as the time from randomization to the first documentation of a 10-point increase from baseline in EORTC QLQ-C30 fatigue scale. EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The symptom scale (fatigue) was scored on a 4-point scale that ranged from "not at all" to "very much". Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher symptom severity). KM method was used to estimate median time to deterioration for each treatment arm.
Time Frame: Up to approximately 34 months
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
months | 1.4 [1.2 to 2.8] | 1.8 [1.5 to 2.8]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.62 to 1.17]

14. Secondary Outcome: Stage 2: Time to Deterioration in Lymphoma Symptoms as Measured by the Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Lymphoma Subscale (FACT-Lym LymS)
Description: Time to deterioration was defined as the time from randomization to the first documentation of a >3-point decrease from baseline in FACT-Lym LymS. The FACT-Lym subscale has 4 domains: physical well-being, social/family well-being, emotional well-being, functional well-being and lymphoma-specific subscale (LymS). The FACT-Lym LYMS consists of common lymphoma disease and/or treatment-related symptoms (e.g., pain, fever, swelling, night sweats, insomnia, itching, weight loss, fatigue, and loss of appetite). FACT-Lym LYMS contains 15 items scored from 0-4, where 0="Not at all" and 4="very much". Scale score range is from 0 to 60. Higher score indicates better quality of life. KM method was used to estimate the median time to deterioration for each treatment arm.
Time Frame: Up to approximately 34 months
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
months | 2.5 [1.4 to 3.2] | 4.6 [2.9 to 7.9]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.45 to 0.91]

15. Secondary Outcome: Stage 2: Change From Baseline in Physical Functioning as Measured by EORTC QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The functioning items were scored on a 4-point scale that ranged from "not at all" to "very much". Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher physical functioning).
Time Frame: Baseline, Day 1 of Cycle 2, 3, 5 and 7 (Cycle length= 21 days), end of treatment, long-term follow-up visits every two months (up to approximately 34 months)
Population: ITT population included all randomized participants. Number analyzed is the number of participants with data available for analysis at the specified timepoint. Participants may have been lost to follow-up/did not complete the specified visit during the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
score on a scale
  Baseline: number analyzed (Participants) | 124 | 127
  Baseline | 65.65 (22.83) | 71.08 (25.09)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 99 | 120
  Change at Cycle 2 Day 1 | -0.88 (16.60) | 0.94 (16.74)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 79 | 111
  Change at Cycle 3 Day 1 | -1.10 (19.81) | 2.16 (19.57)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 47 | 87
  Change at Cycle 5 Day 1 | 1.28 (17.00) | 2.68 (20.65)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 34 | 69
  Change at Cycle 7 Day 1 | -1.76 (18.37) | 0.87 (20.39)
  Change at End of Treatment: number analyzed (Participants) | 86 | 101
  Change at End of Treatment | -4.65 (19.00) | -3.70 (22.56)
  Change at Long-term Follow-up 01: number analyzed (Participants) | 22 | 50
  Change at Long-term Follow-up 01 | 0.91 (19.66) | -0.80 (20.10)
  Change at Long-term Follow-up 02: number analyzed (Participants) | 19 | 38
  Change at Long-term Follow-up 02 | 10.53 (17.54) | 2.28 (20.11)
  Change at Long-term Follow-up 03: number analyzed (Participants) | 14 | 39
  Change at Long-term Follow-up 03 | 4.29 (19.50) | 0.17 (18.51)
  Change at Long-term Follow-up 04: number analyzed (Participants) | 13 | 31
  Change at Long-term Follow-up 04 | 6.67 (15.87) | 0.65 (14.54)
  Change at Long-term Follow-up 05: number analyzed (Participants) | 11 | 29
  Change at Long-term Follow-up 05 | 7.88 (19.28) | -2.53 (18.89)
  Change at Long-term Follow-up 06: number analyzed (Participants) | 10 | 26
  Change at Long-term Follow-up 06 | 10.00 (15.48) | 1.54 (16.79)
  Change at Long-term Follow-up 07: number analyzed (Participants) | 8 | 17
  Change at Long-term Follow-up 07 | 9.17 (17.43) | 6.67 (17.95)
  Change at Long-term Follow-up 08: number analyzed (Participants) | 6 | 11
  Change at Long-term Follow-up 08 | 14.44 (21.26) | 5.45 (16.01)
  Change at Long-term Follow-up 09: number analyzed (Participants) | 6 | 11
  Change at Long-term Follow-up 09 | 16.67 (17.26) | 8.48 (19.57)
  Change at Long-term Follow-up 10: number analyzed (Participants) | 5 | 5
  Change at Long-term Follow-up 10 | 18.67 (18.50) | 5.33 (19.66)
  Change at Long-term Follow-up 11: number analyzed (Participants) | 4 | 4
  Change at Long-term Follow-up 11 | 5.00 (11.39) | 11.67 (15.75)
  Change at Long-term Follow-up 12: number analyzed (Participants) | 3 | 2
  Change at Long-term Follow-up 12 | 13.33 (11.55) | 16.67 (23.57)
  Change at Long-term Follow-up 13: number analyzed (Participants) | 1 | 2
  Change at Long-term Follow-up 13 | 6.67 (NA) — The standard deviation was not estimable for a single participant. | 16.67 (23.57)
  Change at Long-term Follow-up 14: number analyzed (Participants) | 0 | 1
  Change at Long-term Follow-up 14 |  | 33.33 (NA) — The standard deviation was not estimable for a single participant.

16. Secondary Outcome: Stage 2: Change From Baseline in Fatigue Scale as Measured by EORTC QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The symptom scale (fatigue) were scored on a 4-point scale that ranged from "not at all" to "very much". Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher symptom severity). A positive change from baseline indicates an improvement.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 5 and 7 (Cycle length= 21 days), end of treatment, long-term follow-up visits every two months (up to approximately 34 months)
Population: ITT population included all randomized participants. Number analyzed is the number of participants with data available for analysis at the specified time point. Participants may have been lost to follow-up/did not complete the specified visit during the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
score on a scale
  Baseline: number analyzed (Participants) | 124 | 127
  Baseline | 34.99 (25.00) | 35.13 (28.01)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 99 | 119
  Change at Cycle 2 Day 1 | 2.81 (25.16) | 2.57 (20.30)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 79 | 111
  Change at Cycle 3 Day 1 | 2.04 (23.08) | 0.05 (24.39)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 47 | 87
  Change at Cycle 5 Day 1 | 4.26 (25.44) | -0.45 (24.88)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 34 | 69
  Change at Cycle 7 Day 1 | 4.90 (17.56) | 0.48 (27.38)
  Change at End of Treatment: number analyzed (Participants) | 86 | 101
  Change at End of Treatment | 7.43 (26.70) | 6.99 (28.87)
  Change at Long-term Follow-up 01: number analyzed (Participants) | 22 | 50
  Change at Long-term Follow-up 01 | 3.03 (18.84) | -0.67 (23.37)
  Change at Long-term Follow-up 02: number analyzed (Participants) | 19 | 38
  Change at Long-term Follow-up 02 | -8.77 (15.96) | -4.97 (19.96)
  Change at Long-term Follow-up 03: number analyzed (Participants) | 14 | 39
  Change at Long-term Follow-up 03 | 1.59 (24.60) | -6.27 (18.52)
  Change at Long-term Follow-up 04: number analyzed (Participants) | 13 | 31
  Change at Long-term Follow-up 04 | -1.71 (17.48) | -9.68 (18.97)
  Change at Long-term Follow-up 05: number analyzed (Participants) | 11 | 29
  Change at Long-term Follow-up 05 | 0.00 (24.34) | -7.66 (21.23)
  Change at Long-term Follow-up 06: number analyzed (Participants) | 10 | 26
  Change at Long-term Follow-up 06 | 0.00 (25.66) | -7.26 (12.94)
  Change at Long-term Follow-up 07: number analyzed (Participants) | 8 | 17
  Change at Long-term Follow-up 07 | 8.33 (17.57) | -8.50 (16.91)
  Change at Long-term Follow-up 08: number analyzed (Participants) | 6 | 11
  Change at Long-term Follow-up 08 | 0.00 (17.21) | -10.10 (12.62)
  Change at Long-term Follow-up 09: number analyzed (Participants) | 6 | 11
  Change at Long-term Follow-up 09 | 0.00 (23.31) | -12.12 (16.82)
  Change at Long-term Follow-up 10: number analyzed (Participants) | 5 | 5
  Change at Long-term Follow-up 10 | 8.89 (19.88) | -2.22 (4.97)
  Change at Long-term Follow-up 11: number analyzed (Participants) | 4 | 4
  Change at Long-term Follow-up 11 | 11.11 (12.83) | -8.33 (16.67)
  Change at Long-term Follow-up 12: number analyzed (Participants) | 3 | 2
  Change at Long-term Follow-up 12 | 0.00 (19.24) | -11.11 (15.71)
  Change at Long-term Follow-up 13: number analyzed (Participants) | 1 | 2
  Change at Long-term Follow-up 13 | 22.22 (NA) — The standard deviation was not estimable for a single participant. | -11.11 (15.71)
  Change at Long-term Follow-up 14: number analyzed (Participants) | 0 | 1
  Change at Long-term Follow-up 14 |  | -22.22 (NA) — The standard deviation was not estimable for a single participant.

17. Secondary Outcome: Stage 2: Change From Baseline in FACT-Lym LYMS Scores
Description: The FACT-Lym subscale has 4 domains: physical well-being, social/family well-being, emotional well-being, functional well-being and lymphoma-specific subscale (LymS). The FACT-Lym LYMS consists of common lymphoma disease and/or treatment-related symptoms (e.g., pain, fever, swelling, night sweats, insomnia, itching, weight loss, fatigue, and loss of appetite). FACT-Lym LYMS contains 15 items scored from 0-4, where 0="Not at all" and 4="very much". Scale score range is from 0 to 60. Higher score indicates better quality of life. A positive change from baseline indicates an improvement.
Time Frame: as for outcome 15
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
score on a scale
  Baseline: number analyzed (Participants) | 120 | 126
  Baseline | 41.73 (10.88) | 42.49 (10.94)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 98 | 120
  Change at Cycle 2 Day 1 | 0.49 (9.37) | 2.12 (8.38)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 77 | 112
  Change at Cycle 3 Day 1 | 1.71 (8.17) | 2.66 (9.22)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 45 | 87
  Change at Cycle 5 Day 1 | 1.95 (8.15) | 3.53 (8.10)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 34 | 69
  Change at Cycle 7 Day 1 | 0.32 (8.23) | 2.69 (10.45)
  Change at End of Treatment: number analyzed (Participants) | 83 | 100
  Change at End of Treatment | -0.71 (10.34) | 2.34 (11.09)
  Change at Long-term Follow-up 01: number analyzed (Participants) | 21 | 49
  Change at Long-term Follow-up 01 | 0.14 (13.10) | 2.88 (10.03)
  Change at Long-term Follow-up 02: number analyzed (Participants) | 18 | 38
  Change at Long-term Follow-up 02 | 5.22 (9.28) | 5.32 (8.15)
  Change at Long-term Follow-up 03: number analyzed (Participants) | 13 | 39
  Change at Long-term Follow-up 03 | 4.08 (7.31) | 3.90 (7.32)
  Change at Long-term Follow-up 04: number analyzed (Participants) | 12 | 31
  Change at Long-term Follow-up 04 | 6.00 (6.18) | 4.29 (6.47)
  Change at Long-term Follow-up 05: number analyzed (Participants) | 10 | 28
  Change at Long-term Follow-up 05 | 6.00 (9.56) | 4.07 (6.87)
  Change at Long-term Follow-up 06: number analyzed (Participants) | 9 | 27
  Change at Long-term Follow-up 06 | 5.89 (6.75) | 4.15 (6.16)
  Change at Long-term Follow-up 07: number analyzed (Participants) | 7 | 17
  Change at Long-term Follow-up 07 | 5.29 (7.54) | 4.65 (7.56)
  Change at Long-term Follow-up 08: number analyzed (Participants) | 5 | 11
  Change at Long-term Follow-up 08 | 8.00 (4.53) | 5.82 (5.46)
  Change at Long-term Follow-up 09: number analyzed (Participants) | 5 | 11
  Change at Long-term Follow-up 09 | 8.80 (5.81) | 7.82 (6.63)
  Change at Long-term Follow-up 10: number analyzed (Participants) | 4 | 5
  Change at Long-term Follow-up 10 | 7.50 (7.23) | 4.00 (3.32)
  Change at Long-term Follow-up 11: number analyzed (Participants) | 3 | 4
  Change at Long-term Follow-up 11 | 5.67 (7.02) | 6.75 (5.44)
  Change at Long-term Follow-up 12: number analyzed (Participants) | 2 | 2
  Change at Long-term Follow-up 12 | 5.50 (0.71) | 4.50 (4.95)
  Change at Long-term Follow-up 13: number analyzed (Participants) | 1 | 2
  Change at Long-term Follow-up 13 | 13.00 (NA) — The standard deviation was not estimable for a single participant. | 4.00 (4.24)
  Change at Long-term Follow-up 14: number analyzed (Participants) | 0 | 1
  Change at Long-term Follow-up 14 |  | 8.00 (NA) — The standard deviation was not estimable for a single participant.

18. Secondary Outcome: Stage 2: Change From Baseline in Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity 12-Item (FACT/GOG-NTX-12) Scores
Description: The FACT/GOG-NTX scale provides a targeted assessment of symptoms of peripheral neuropathy, including sensory, motor, and auditory problems and cold sensitivity. It contains 12 items scored from 0-4, where 0="Not at all" and 4="very much". Scores are summed for a range of 12-44, with lower scores indicating more severe neurotoxicity. Participants completed assessments until progression or non-protocol-specified anti-lymphoma treatment (NALT). Only records on or before the first NALT were summarized.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7 and 8 (Cycle length= 21 days), end of treatment, long-term follow-up visits every two months (up to approximately 34 months)
Population: Safety run-in population included all participants who received any amount of any study drug during safety run-in stage. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints. Participants may have been lost to follow-up/did not complete the specified visit during the study.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 125 | 128
score on scale
  Baseline: number analyzed (Participants) | 124 | 127
  Baseline | 40.67 (6.70) | 40.37 (8.32)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 100 | 121
  Change at Cycle 2 Day 1 | -1.56 (5.60) | -0.54 (6.87)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 80 | 113
  Change at Cycle 3 Day 1 | -1.35 (4.91) | -0.20 (8.01)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 70 | 106
  Change at Cycle 4 Day 1 | -2.44 (6.82) | -0.78 (7.58)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 46 | 87
  Change at Cycle 5 Day 1 | -2.35 (4.54) | -1.68 (7.95)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 41 | 76
  Change at Cycle 6 Day 1 | -2.02 (5.47) | -3.48 (8.92)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 35 | 69
  Change at Cycle 7 Day 1 | -2.00 (4.77) | -4.25 (9.97)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 29 | 62
  Change at Cycle 8 Day 1 | -3.62 (4.95) | -5.08 (10.41)
  Change at End of Treatment: number analyzed (Participants) | 85 | 100
  Change at End of Treatment | -3.80 (7.65) | -5.96 (11.05)
  Change at Long-term Follow-up 01: number analyzed (Participants) | 22 | 50
  Change at Long-term Follow-up 01 | -4.91 (9.11) | -9.50 (11.00)
  Change at Long-term Follow-up 02: number analyzed (Participants) | 19 | 38
  Change at Long-term Follow-up 02 | -3.77 (7.00) | -6.86 (7.75)
  Change at Long-term Follow-up 03: number analyzed (Participants) | 15 | 39
  Change at Long-term Follow-up 03 | -4.73 (7.22) | -7.73 (7.04)
  Change at Long-term Follow-up 04: number analyzed (Participants) | 13 | 31
  Change at Long-term Follow-up 04 | -0.85 (6.35) | -5.18 (5.96)
  Change at Long-term Follow-up 05: number analyzed (Participants) | 11 | 29
  Change at Long-term Follow-up 05 | -1.55 (3.91) | -4.92 (5.85)
  Change at Long-term Follow-up 06: number analyzed (Participants) | 10 | 27
  Change at Long-term Follow-up 06 | -1.20 (5.22) | -4.58 (6.79)
  Change at Long-term Follow-up 07: number analyzed (Participants) | 8 | 17
  Change at Long-term Follow-up 07 | -3.00 (6.55) | -3.62 (6.18)
  Change at Long-term Follow-up 08: number analyzed (Participants) | 6 | 11
  Change at Long-term Follow-up 08 | 0.83 (5.71) | -3.05 (7.02)
  Change at Long-term Follow-up 09: number analyzed (Participants) | 6 | 10
  Change at Long-term Follow-up 09 | 0.83 (5.56) | -4.20 (4.42)
  Change at Long-term Follow-up 10: number analyzed (Participants) | 5 | 5
  Change at Long-term Follow-up 10 | 1.20 (7.40) | -4.60 (6.02)
  Change at Long-term Follow-up 11: number analyzed (Participants) | 4 | 4
  Change at Long-term Follow-up 11 | -1.50 (4.80) | -1.50 (1.91)
  Change at Long-term Follow-up 12: number analyzed (Participants) | 3 | 2
  Change at Long-term Follow-up 12 | -0.33 (4.16) | -1.50 (0.71)
  Change at Long-term Follow-up 13: number analyzed (Participants) | 1 | 2
  Change at Long-term Follow-up 13 | -5.00 (NA) — The standard deviation was not estimable for a single participant. | -2.00 (0.00)
  Change at Long-term Follow-up 14: number analyzed (Participants) | 0 | 1
  Change at Long-term Follow-up 14 |  | 39.00 (NA) — The standard deviation was not estimable for a single participant.
  Change at Long-term Follow-up 16: number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Stage 2: Percentage of Participants With Clinically Meaningful Improvement in EORTC QLQ-C30 Physical Functioning Scale
Description: EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The functioning items were scored on a 4-point scale that ranged from "not at all" to "very much". Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher functioning). Clinically meaningful improvement was defined as a participant with at least a 7 point scale score increase.
Time Frame: Up to approximately 34 months
Population: ITT population included all randomized participants in Stage 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
percentage of participants | 31.0 [23.02 to 39.80] | 41.1 [32.50 to 50.09]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Difference in Response Rate = 10.13, 95% CI 2-sided [-2.37 to 22.63]

20. Secondary Outcome: Stage 2: Percentage of Participants With Clinically Meaningful Improvement in EORTC QLQ-C30 Fatigue Scale
Description: EORTC QLQ-C30 consists of 30 questions assessing five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), GHS/QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The symptom items were scored on a 4-point scale that ranged from "not at all" to "very much". Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher symptom severity). Clinically meaningful improvement was defined as a participant with at least a 9 point scale score decrease.
Time Frame: Up to approximately 34 months
Population: ITT population included all randomized participants in Stage 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
percentage of participants | 46.0 [37.12 to 55.14] | 55.8 [46.81 to 64.55]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Difference in Response Rate = 9.78, 95% CI 2-sided [-3.22 to 22.78]

21. Secondary Outcome: Stage 2: Percentage of Participants With Clinically Meaningful Improvement in FACT-Lym LYMS
Description: The FACT-Lym subscale has 4 domains: physical well-being, social/family well-being, emotional well-being, functional well-being and lymphoma-specific subscale (LymS). The FACT-Lym LYMS consists of common lymphoma disease and/or treatment-related symptoms (e.g., pain, fever, swelling, night sweats, insomnia, itching, weight loss, fatigue, and loss of appetite). FACT-Lym LYMS contains 15 items scored from 0-4, where 0="Not at all" and 4="very much". Scale score range is from 0 to 60. Higher score indicates better quality of life. Clinically meaningful improvement was defined as a 3-point increase from baseline.
Time Frame: Up to approximately 34 months
Population: ITT population included all randomized participants in Stage 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 126 | 129
percentage of participants | 48.4 [39.42 to 57.48] | 66.7 [57.83 to 74.72]
Statistical Analysis 1: Comparison: Stage 2: R-GemOx vs Stage 2: Pola-R-GemOx; Test type: Superiority; Difference in Response Rate = 18.25, 95% CI 2-sided [5.54 to 30.97]

22. Secondary Outcome: Stage 2: Number of Participants With AEs
Description: as for outcome 1
Time Frame: From treatment initiation until 90 days after the last dose of study drug or initiation of NALT (approximately 10.6 months)
Population: Safety-evaluable population included all participants who received any amount of any study drug (regardless of the stage).
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 125 | 128
Participants | 117 | 125

23. Secondary Outcome: Stage 2: Number of Participants With PN
Description: as for outcome 2
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 125 | 128
Participants | 36 | 73

24. Secondary Outcome: Stage 1 and Stage 2: Number of Participants With Dose Modification for Polatuzumab Vedotin
Description: Dose modifications (interruptions/reductions) were based on physical examination findings, observed toxicities, and laboratory results obtained within 72 hours before study treatment administration. The determination of all dose modifications was made based on the investigator's assessment of ongoing clinical benefit with continuing study treatment. Dosing occurred only when a participant's clinical assessment and laboratory test values were acceptable.
Time Frame: Stage 1: Up to approximately 5.3 months and Stage 2: Up to approximately 7.6 months
Population: Safety population included all participants who received any amount of any study drug (regardless of the stage).
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 128
Participants | 3 | 22

25. Secondary Outcome: Stage 1 and Stage 2: Dose Intensity of Polatuzumab Vedotin
Description: Dose intensity = (total dose actually received divided by the expected total dose)*100. Expected total dose for dose intensity accounting for delay/reduction is based on the expected number of cycles between the first and last exposure of each drug. Percentage of dose intensity accounting for delay/reduction in dose by the participants in each arm is reported here.
Time Frame: Stage 1: Up to approximately 5.3 months and Stage 2: Up to approximately 7.6 months
Population: Safety population included all participants who received any amount of any study drug (regardless of the stage).
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 15 | 128
percentage of dose | 93.60 (11.23) | 92.81 (10.33)

26. Secondary Outcome: Stage 1: OS
Description: OS was defined as the time from randomization to the death from any cause during the study. Participants who were not reported as having died at the time of analysis were censored at the date when they were last known to be alive. Participants who did not have post-baseline information were censored at the date of randomization. KM method was used to estimate median OS for each treatment arm.
Time Frame: From randomization to the death (up to approximately 34 months)
Population: Safety run-in population included all participants who received any amount of any study drug during safety run-in stage.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: Pola-R-GemOx
Number analyzed (Participants) | 15
months | 12.6 [11.4 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

27. Secondary Outcome: Stage 1 and Stage 2: Percentage of Participants With Anti-drug Antibodies (ADAs) to Polatuzumab Vedotin
Description: Treatment emergent ADA-positive participants after drug administration were determined for participants exposed to polatuzumab vedotin. Participants positive for treatment emergent ADA were defined as the number of post-baseline evaluable participants determined to have treatment-induced ADA or treatment-enhanced ADA during the study period. Treatment-induced ADA = a participant with negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result. Percentages are rounded off.
Time Frame: Up to approximately 34 months
Population: Immunogenicity-evaluable population included all participants who received at least one dose of polatuzumab vedotin with at least one evaluable post-baseline ADA sample.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: Pola-R-GemOx
Number analyzed (Participants) | 12 | 117
percentage of participants | 0 | 2.6

ADVERSE EVENTS:
Time Frame: AEs and SAEs: From treatment initiation until 90 days after the last dose of study drug or initiation of NALT (approximately 8.3 months for Stage 1 and 10.6 months for Stage 2). All-cause Mortality: Up to approximately 34 months
Description: Safety population included all participants who received any amount of any study drug (regardless of the stage). 1 participant in each Pola-R-GemOx arm and R-GemOx arm of Stage 2 did not receive any treatment and were excluded from the safety population.
Groups:
- Stage 1: Pola-R-GemOx: Participants received rituximab, 375 milligrams mg/m^2, IV, followed by polatuzumab vedotin, 1.8 mg/kg, IV on Day 1 of each 21-day cycle. Participants also received gemcitabine, 1000 mg/m^2, IV followed by oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
- Pola-R-GemOx - Pooled: All participants who received rituximab, 375 mg/m^2, IV, followed by polatuzumab vedotin, 1.8 mg/kg, IV on Day 1 of each 21-day cycle either during safety run-in or RCT stage, were included in this arm. Participants also received gemcitabine, 1000 mg/m^2, IV followed by oxaliplatin 100 mg/m^2, IV on Day 2 of each 21-day cycle for up to 8 cycles.
Arm/Group | Stage 1: Pola-R-GemOx | Stage 2: R-GemOx | Stage 2: Pola-R-GemOx | Pola-R-GemOx - Pooled
All-Cause Mortality (participants affected / at risk) | 9/15 | 83/125 | 68/128 | 77/143
Serious Adverse Events (participants affected / at risk) | 2/15 | 39/125 | 49/128 | 51/143
Other Adverse Events (participants affected / at risk) | 14/15 | 111/125 | 119/128 | 133/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Pola-R-GemOx (N=15) | Stage 2: R-GemOx (N=125) | Stage 2: Pola-R-GemOx (N=128) | Pola-R-GemOx - Pooled (N=143)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 2 (2) | 3 (3)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (7) | 6 (7)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 2 (3) | 2 (3)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 8 (8) | 8 (8)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 9 (10) | 9 (10)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematological infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection in an immunocompromised host (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Meningitis listeria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 5 (5) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (5) | 1 (2) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 2 (6) | 2 (6)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (3) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Pola-R-GemOx (N=15) | Stage 2: R-GemOx (N=125) | Stage 2: Pola-R-GemOx (N=128) | Pola-R-GemOx - Pooled (N=143)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 32 (54) | 48 (101) | 50 (103)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 2 (2) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 10 (14) | 4 (14) | 4 (14)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 22 (49) | 24 (71) | 27 (77)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (8) | 22 (45) | 30 (96) | 34 (104)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 7 (7) | 8 (9) | 8 (9)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 12 (15) | 17 (19) | 22 (25)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 26 (35) | 47 (87) | 51 (94)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 42 (72) | 50 (128) | 54 (133)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 35 (60) | 34 (62) | 36 (65)
Asthenia (General disorders) | 1 (1) | 4 (4) | 11 (13) | 12 (14)
Chest pain (General disorders) | 1 (1) | 2 (3) | 4 (5) | 5 (6)
Chills (General disorders) | 1 (1) | 2 (2) | 5 (5) | 6 (6)
Device related thrombosis (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 5 (5) | 10 (12) | 13 (13) | 18 (18)
Infusion site extravasation (General disorders) | 2 (2) | 3 (4) | 1 (1) | 3 (3)
Malaise (General disorders) | 0 (0) | 6 (15) | 11 (21) | 11 (21)
Oedema peripheral (General disorders) | 1 (1) | 5 (5) | 6 (6) | 7 (7)
Pyrexia (General disorders) | 4 (4) | 20 (24) | 18 (24) | 22 (28)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 14 (15) | 15 (16) | 15 (16)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 19 (24) | 29 (56) | 31 (58)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 18 (24) | 31 (61) | 33 (63)
Blood creatinine increased (Investigations) | 1 (1) | 5 (10) | 7 (15) | 8 (16)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 9 (9) | 10 (11) | 10 (11)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (11) | 13 (30) | 13 (30)
Neutrophil count decreased (Investigations) | 0 (0) | 27 (60) | 29 (98) | 29 (98)
Platelet count decreased (Investigations) | 0 (0) | 27 (57) | 38 (115) | 38 (115)
Weight decreased (Investigations) | 2 (2) | 10 (10) | 15 (16) | 17 (18)
White blood cell count decreased (Investigations) | 0 (0) | 28 (53) | 25 (84) | 25 (84)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 18 (27) | 29 (60) | 31 (62)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 8 (14) | 8 (14)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (7) | 3 (4) | 4 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (9) | 8 (12) | 8 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 9 (11) | 14 (33) | 17 (36)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 7 (20) | 8 (21)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (6) | 4 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 7 (8) | 6 (6) | 6 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 1 (2) | 7 (8) | 12 (15) | 13 (17)
Neuropathy peripheral (Nervous system disorders) | 4 (13) | 25 (37) | 56 (94) | 60 (107)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 8 (8) | 10 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 6 (15) | 8 (11) | 10 (13)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 11 (11) | 16 (17) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 6 (6) | 10 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (5) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (5) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (11) | 5 (5) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 3 (4) | 9 (16) | 10 (16) | 13 (20)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1) | 3 (8) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT04182204/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04182204/SAP_001.pdf